CLINICAL TRIAL: NCT01978691
Title: The Effect of Separate or Combined Supplementation of Probiotic (Bifidobacterium Lactis B420) and Polydextrose on Body Fat Mass
Brief Title: The Effect of a Bifidobacterium and Polydextrose on Body Fat Mass
Acronym: MetSProb
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Danisco (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SMR-2782
Record Dates: First submitted 2013-11-01; First posted 2013-11-07 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Obesity; Hyperglycemia; Insulin Resistance
Keywords: Obesity; Blood glucose; Waist circumference; Lipid metabolism; Probiotics; Prebiotics; Dietary supplements; Endotoxemia
MeSH Terms: conditions — Obesity; Hyperglycemia; Insulin Resistance; Endotoxemia | interventions — 20-aldehyde leukotriene B4; polydextrose; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Probiotic (Active Comparator): Bifidobacterium animalis ssp. lactis 420 (10^10 colony-forming units (CFU)/day in 12 g of microcrystalline cellulose), once per day for six months in a sachet mixed into a smoothie drink
  Interventions: Dietary Supplement: Bifidobacterium animalis ssp. lactis 420
- Prebiotic (Active Comparator): Polydextrose, 12 g once per day for six months in a sachet mixed into a smoothie drink
  Interventions: Dietary Supplement: Polydextrose
- Synbiotic (Active Comparator): B. lactis 420 (10^10 CFU/day) in 12 g of polydextrose, once per day for six months in a sachet to be mixed into a smoothie drink
  Interventions: Dietary Supplement: Bifidobacterium animalis ssp. lactis 420; Dietary Supplement: Polydextrose
- Control (Placebo Comparator): 12 g of microcrystalline cellulose once per day for six months in a sachet to be mixed into a smoothie drink
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Bifidobacterium animalis ssp. lactis 420 — Studied as a probiotic bacteria
  Other Names: B420
  Arms: Probiotic; Synbiotic
Dietary Supplement: Polydextrose — Studied as a prebiotic
  Other Names: Litesse; Litesse Ultra
  Arms: Prebiotic; Synbiotic
Other: Placebo — Control
  Other Names: Microcrystalline cellulose
  Arms: Control

SUMMARY:
Obesity is a major problem worldwide, and it is related to abnormalities in glucose and lipid metabolism. The purpose of this study is to investigate the effect of a dietary supplement containing probiotic (Bifidobacterium animalis ssp. lactis 420) and/or prebiotic (Litesse) on change in body fat mass in a double-blind, randomized, placebo-controlled intervention trial. The supplement is ingested once per day for the duration of six months, and participants will attend a follow-up visit one month after the end of the intervention. The study will enroll 232 participants (58 per study arm) in four research centers in southern Finland.

DETAILED DESCRIPTION:
Obesity is a major problem worldwide, and it is related to abnormalities in glucose and lipid metabolism. Preclinical studies have shown that weight gain and insulin resistance may be prevented by oral administration of the probiotic Bifidobacterium animalis ssp. lactis 420. Furthermore, the prebiotic polydextrose has shown efficacy on satiety in clinical settings. The purpose of this study is to investigate the effects of these products, individually and combined, on change in body fat mass in a double-blind, randomized, placebo-controlled intervention trial. The study is conducted at four research clinics in southern Finland. The supplement is provided in a sachet, mixed into a fruit smoothie and ingested once per day for the duration of six months. One month from the end of the intervention participants will attend a follow-up visit. The study will enroll 232 participants, who will be randomized into blocks using a computerized procedure.

After the screening visit, there will be seven study visits (once per month) and one follow-up visit. Visits at months 0, 2, 4, 6 and follow-up are clinic visits, and visits at months 1, 3 and 5 are phone contacts to check compliance and any adverse events.

Clinic visits include the following measurements and samples:

* weight
* blood pressure and heart rate
* blood samples
* returning of food diaries (only during intervention)
* returning of exercise questionnaires and food choice questionnaires (only beginning and end of treatment)
* returning of fecal samples, taken at home by participant
* DXA for body composition analysis
* hip and waist circumference
* brief physical examination (only beginning and end of treatment)
* recording of adverse events and concomitant medication

For compliance check, unused sachets are returned to the clinic and counted. At the follow-up visit participants will receive guidance on exercise and a healthy diet.

The primary variable of this study is relative change from baseline to end-of-treatment in body fat mass. Comparisons between each of the active groups against the placebo group will be performed if the global P-value is significant. Secondary variables will be analyzed in a similar fashion. The relative and absolute changes in body fat mass will also be analyzed. To explore the mechanism of potential treatment benefits, post-hoc responder analyses may optionally be performed. Also, correlations between the response variables may be examined in exploratory analyses. Post-hoc analyses may be conducted to compare e.g. different time points or to analyze differences from end-of-treatment to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 28.0-34.9
* Waist to hip ratio: males ≥0.88, females ≥0.83
* Age 18-65 years
* Signed informed consent
* Available for all study visits and phone calls
* Follows a regular diet that is in agreement with the national dietary recommendations

Exclusion Criteria:

* Diagnosed type 1 or type 2 diabetes (i.e. fasting plasma glucose ≥ 7 mmol/l and HbA1C ≥ 6.5%)
* Use of medication for diabetes, dyslipidemia or hypertension
* Use of laxatives or fiber supplements in the past 6 weeks
* History of diagnosed coronary heart disease, other significant cardiovascular disease or artificial heart valve
* History of chronic active inflammatory disorders
* History of bariatric surgery
* Use of anti-obesity drugs in the last 3 months
* Use of anticoagulants
* Regular use of non-steroidal anti-inflammatory drugs, systemic or inhaled corticosteroids, or systemic immunomodulatory drugs
* Recent (last 2 months) or ongoing antibiotic use
* Immunosuppression or ongoing therapy causing immunosuppression
* Use of probiotics more than once a week during the previous 6 weeks
* Use of vitamin D supplementation:

  1. > 50 - <100 µg/day during the previous 2 weeks
  2. ≥ 100 - <150 µg/day during the previous 2 months
  3. ≥150 µg/day or above during the previous 12 months
* Active or recent (last 3 months) participation in a weight loss program or weight change (increase or loss) of 3 kg during the past 3 months
* Pregnant or planning pregnancy within 6 months or breastfeeding women
* Participation in a clinical trial with an investigational product or drug within 60 days prior to screening
* Likeliness to be noncompliant with the protocol
* Drug or alcohol abuse
* Allergy to any of the ingredients used in the study
* Other reasons that, in the opinion of the Investigator makes the subject unsuitable for enrolment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Difference in body fat mass from baseline to end-of-treatment (6 months) | From baseline to end of intervention (6 months)
  Measured with dual-energy x-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Change in weight (absolute and relative) | Months 0, 2, 4, 6 and 7 (follow-up)
Change in BMI (absolute and relative) | Months 0, 2, 4, 6 and 7 (follow-up)
Change in lean body mass | Months 0, 2, 4, 6 and 7 (follow-up)
  Total, and in individual regions of the body
Hip Change in waist and/or hip circumference (absolute and relative) | Months 0, 2, 4, 6 and 7 (follow-up)
Change in glycated haemoglobin (HbA1c) in blood | Months 0, 2, 4, 6 and 7 (follow-up)
Change in fasting glucose levels | Months 0, 2, 4, 6 and 7 (follow-up)
Change in fasting insulin levels | Months 0, 2, 4, 6 and 7 (follow-up)
Change in insulin resistance | Months 0, 2, 4, 6 and 7 (follow-up)
  As determined by Homeostasis Model Assessment (HOMA)
Change in inflammatory markers | Months 0, 2, 4, 6 and 7 (follow-up)
  Including high-sensitive C-reactive protein (CRP), Interleukin (IL)-6, Tumor necrosis factor (TNF)-alpha, IL-1beta, cortisol, adiponectin, leptin
Change in lipopolysaccharide (LPS) concentration and soluble CD14 (sCD14) | Months 0, 2, 4, 6 and 7 (follow-up)
Change in LPS/sCD14 ratio | Months 0, 2, 4, 6 and 7 (follow-up)
Change in blood lipids | Months 0, 2, 4, 6 and 7 (follow-up)
  Total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides
Change in blood pressure | Months 0, 2, 4, 6 and 7 (follow-up)
Change in aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT) and gamma-glutamyltransferase | Months 0, 2, 4, 6 and 7 (follow-up)
Change in energy, fat and fiber intake | Months 0, 2, 4, 6 and 7 (follow-up)
Absolute change in body fat mass | Months 0, 2, 4, 6 and 7 (follow-up)
Analytical description of faecal microbiota | Months 0, 2, 4, 6 and 7 (follow-up)
Body fat mass in individual regions of the body | Months 0, 2, 4, 6 and 7 (follow-up)

OTHER OUTCOMES:
The differences between the treatment groups for exploratory variables | Throughout the 6-month study and 1-month follow-up
  Fecal fat and/or energy content, change in plasma and fecal bile acids, plasma oxidated low-density lipoprotein cholesterol, LPS binding protein, Macrophage chemoattractant protein-1, Angiopoietin-like factor 4, Apolipoprotein B-48, Plasminogen activator inhibitor-1, Vascular cell adhesion molecule-1, Intercellular adhesion molecule-1, E-selectin, zonulin, blood microbiota

CONTACTS AND LOCATIONS:
Overall Officials: Aila Rissanen, MD, Principal Investigator — HYKS-instituutti Oy
Locations (4):
- Finland (4):
  - VL-Medi, Helsinki
  - Kerava healthcare center, Kerava
  - FinnMedi Oy, Tampere
  - CRST - Clinical Research Services Turku, Turku

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Amar J, Chabo C, Waget A, Klopp P, Vachoux C, Bermudez-Humaran LG, Smirnova N, Berge M, Sulpice T, Lahtinen S, Ouwehand A, Langella P, Rautonen N, Sansonetti PJ, Burcelin R. Intestinal mucosal adherence and translocation of commensal bacteria at the early onset of type 2 diabetes: molecular mechanisms and probiotic treatment. EMBO Mol Med. 2011 Sep;3(9):559-72. doi: 10.1002/emmm.201100159. Epub 2011 Aug 3. PMID 21735552
- [Derived] Hibberd AA, Yde CC, Ziegler ML, Honore AH, Saarinen MT, Lahtinen S, Stahl B, Jensen HM, Stenman LK. Probiotic or synbiotic alters the gut microbiota and metabolism in a randomised controlled trial of weight management in overweight adults. Benef Microbes. 2019 Mar 13;10(2):121-135. doi: 10.3920/BM2018.0028. Epub 2018 Dec 10. PMID 30525950
- [Derived] Stenman LK, Lehtinen MJ, Meland N, Christensen JE, Yeung N, Saarinen MT, Courtney M, Burcelin R, Lahdeaho ML, Linros J, Apter D, Scheinin M, Kloster Smerud H, Rissanen A, Lahtinen S. Probiotic With or Without Fiber Controls Body Fat Mass, Associated With Serum Zonulin, in Overweight and Obese Adults-Randomized Controlled Trial. EBioMedicine. 2016 Nov;13:190-200. doi: 10.1016/j.ebiom.2016.10.036. Epub 2016 Oct 26. PMID 27810310